CLINICAL TRIAL: NCT03273166
Title: Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance During Hemodilution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-18788
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Healthy
MeSH Terms: interventions — Hemodilution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- INVSENSOR00001 sensor (Experimental): This is a nonrandomized single arm study wherein all subjects are enrolled into the experimental arm and receive both the INVSENSOR00001 sensor and the control sensor simultaneously on different fingers.
  Interventions: Device: INVSENSOR00001; Device: Control SpHb sensor; Procedure: Hemodilution

INTERVENTIONS:
Device: INVSENSOR00001 — This is a non-randomized single arm study wherein all subjects are enrolled into the experimental arm and receive both the INVSENSOR00001 sensor and the control sensor simultaneously on different fingers.
Device: Control SpHb sensor — This is a non-randomized single arm study wherein all subjects are enrolled into the experimental arm and receive both the INVSENSOR00001 sensor and the control sensor simultaneously on different fingers.
Procedure: Hemodilution — This is a non-randomized single arm study wherein all subjects are enrolled into the experimental arm and receive both the INVSENSOR00001 sensor and the control sensor simultaneously on different fingers while undergoing a hemodilution procedure.

SUMMARY:
This study involves comparison of the performance of two SpHb sensors in subjects that undergo a hemodilution procedure. The sensors' performance will be assessed by comparison of the measured hemoglobin values against reference values obtained by a laboratory hematology analyzer. Blood samples will be collected from healthy volunteers who undergo a hemodilution procedure wherein blood is repeatedly sampled as the concentration of hemoglobin is reduced by administering intravenous fluids to the volunteer in a controlled manner.

ELIGIBILITY:
Inclusion Criteria:

* Competent adults between the ages of 18 and 50 years of age
* Must weigh a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall
* BMI ≤ 35 unless the physician determines that a higher BMI is not due to morbid obesity, to safeguard subject safety during hemodilution
* Must have a hemoglobin value ≥ 11 g/dL at time of screening, to safeguard subject safety during hemodilution
* Baseline heart rate between 45 bpm and 85 bpm
* CO value less than 2.0% FCOHb
* Physical status of ASA I or II (American Society of Anesthesiology Class I; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) The ASA definition strictly applies to the systemic disease portion of the classification
* Systolic BP less than or equal to 140 mmHg and Diastolic BP less than or equal to 90 mmHg
* Able to read and communicate in English

Exclusion Criteria:

* Pregnancy or positive hCG test
* Smokers (including e-cigarette users)
* Subject has known drug or alcohol abuse. Subjects who uses recreational drugs
* Subject has experienced a concussion or head injury with loss of consciousness within the last year
* Any chronic bleeding disorders (i.e. hemophilia)
* Any history of a stroke, myocardial infarction, or seizures
* Any cancer or history of cancer (not including skin cancer)
* Chronic neurological diseases (i.e. multiple sclerosis, Huntington's Disease)
* Any cardiac dysrhythmias (i.e. atrial fibrillation)(without physicians clearance)
* Subject has known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder) that interferes with the subject's level of consciousness
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome
* Subjects who have/are currently taking anticoagulant medication
* Subjects who have taken opioid pain medication within 24 hours of start of study
* Subjects who do not understand the study and the risks
* Subjects having either signs or history of peripheral ischemia
* Subjects who have had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, plastic surgery, major ENT surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery
* Subjects that have symptoms of congestion, head colds, flu, or other illnesses
* Subjects with claustrophobia, or generalized anxiety disorder
* Subjects who have been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months
* Subjects with chronic unresolved asthma, lung disease and respiratory disease
* Subjects with allergies to lidocaine, latex, adhesives, or plastic
* Subjects with heart conditions, insulin-dependent diabetes or uncontrolled hypertension
* Subjects who have given vaginal delivery, had a pregnancy terminated, a miscarriage with hospitalization or had a c-section within the last 6 months
* Subjects who intend on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours following a study involving an arterial blood draw and/or arterial line placement
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fingers were not randomized to the two interventions. All participants received both interventions in the exact same manner.
Groups:
- INVSENSOR00001: All subjects consented are enrolled into the test group and will receive the INVSENSOR00001 and the control sensor simultaneously on different fingers.
Period: Overall Study
Arm/Group | INVSENSOR00001
Started | 82
Completed | 51
Not Completed | 31
Not completed — Withdrawn prior to Completion | 31

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00001
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity, Customized: Caucasian | 17
  Race/Ethnicity, Customized: Hispanic | 16
  Race/Ethnicity, Customized: Asian or Pacific Islander | 3
  Race/Ethnicity, Customized: Native American | 2
  Race/Ethnicity, Customized: Black or African American | 13
  Race/Ethnicity, Customized: Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Comparison of INVSENSOR00001 and Control SpHb Sensor by ARMS Calculation
Description: Performance of the sensors will be determined by comparing the noninvasive hemoglobin measurement (SpHb) of the pulse oximeter sensors to the hemoglobin value obtained from a reference blood sample and calculating the accuracy root mean square(ARMS) value.
Time Frame: 1-5 hours
Measure: Number; unit: g/dL
Groups:
- Control SpHb Sensor: All subjects consented are enrolled into the test group and will receive the INVSENSOR00001 and the control sensor simultaneously on different fingers.
Arm/Group | INVSENSOR00001 | Control SpHb Sensor
Number analyzed (Participants) | 51 | 51
g/dL | 0.9 | 0.9

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Description: Adverse Events were not collected with respect to the interventions, only on participants as a whole.
Arm/Group | INVSENSOR00001
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 2/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INVSENSOR00001 (N=51)
Dizziness (Injury, poisoning and procedural complications) | 1
Irregular EKG readings (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03273166/Prot_SAP_000.pdf